CLINICAL TRIAL: NCT04515615
Title: A Multi-center, Phase II Study to Evaluate Safety and Efficacy of Adjuvant Chemotherapy With Tegafur Gimeracil Oteracil Potassium Capsule Plus Oxaliplatin and Camrelizumab for Stage III Gastric Cancer (FOCUS-02)
Brief Title: Adjuvant Chemotherapy in Combination With Camrelizumab for Stage III Gastric Cancer (FOCUS-02)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yu jiren (Other)
Responsible Party: Sponsor-Investigator, Yu jiren, Director of gastrointestinal surgery department, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20200046C-R1
Record Dates: First submitted 2020-08-14; First posted 2020-08-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastric Cancer Stage III
Keywords: Gastric cancer; Camrelizumab; Chemotherapy; Phase II
MeSH Terms: conditions — Stomach Neoplasms | interventions — camrelizumab; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab and chemotherapy (Experimental): Participants receive camrelizumab 200 mg intravenously (IV) on the first day (q3w), then oxaliplatin 130 mg/m^2, IV on the first day (q3w), and tegafur gimeracil oteracil potassium capsule 80 mg/m^2 twice daily (BID) by continuous oral administration for 14 days, followed by a recovery period of 7 days. Three weeks as a course of treatment, a total of 8 courses.
  Interventions: Drug: Camrelizumab; Drug: Oxaliplatin; Drug: Tegafur gimeracil oteracil potassium capsule

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab, 200 mg IV for 30-60 min in first day every 3 weeks. Repeated every 21 days. 21 days for a cycle.
  Other Names: SHR-1210
Drug: Oxaliplatin — Oxaliplatin: 130 mg/m^2 IV for 2-6 hour in first day which will be administered at least 30 min after completion of camrelizumab administration, every 3 weeks. Repeated every 21 days, 21 days for a cycle.
Drug: Tegafur gimeracil oteracil potassium capsule — Tegafur gimeracil oteracil potassium capsule: 80 mg/m^2 twice daily (BID) by continuous oral administration for 14 days, followed by a recovery period of 7 days. Repeated every 21 days. 21 days for a cycle.

SUMMARY:
This study is a prospective, single arm, multi-center phase II clinical trial. The primary study objective is to evaluate the safety of tegafur gimeracil oteracil potassium capsule plus oxaliplatin and Camrelizumab as adjuvant therapy in stage III gastric cancer, including the incidences and types of adverse events. The secondary study objective is to observe and evaluate the disease-free survival (DFS), overall survival (OS) and treatment completion rate.

DETAILED DESCRIPTION:
1. Study population: participants with stage III gastric cancer confirmed by postoperative pathology according to American Joint Committee on Cancer (AJCC) / Union for International Cancer Control (UICC) 8th Tumor Node Metastasis (TNM) staging classification.
2. Sample size: single arm design was used in this study and 52 participants were estimated to be enrolled.
3. Research content: In this study, within 4-6 weeks after the completion of the operation, the participants were selected and qualified for this study, and were scheduled to receive 200mg camrelizumab once intravenous infusion on the first day (q3w), then 130mg/m^2 oxaliplatin on the first day (q3w), and tegafur gimeracil oteracil potassium capsule was taken as follow: surface area is less than 1.25, 80mg per day, twice a day; ≥1.25 ~ <1.5, 100mg per day, twice a day; ≥1.5, 120mg per day, twice a day, and oral administration for 1-14 days every 3 weeks. Three weeks as a course of treatment, a total of 8 courses, after treatment, safety visit and survival follow-up will be carried out. A total of 3 years follow-up time is scheduled since the first medication, and the frequency is once every 3-6 months within 2 years, and once every 6-12 months for the third year.
4. Adverse events (AEs) management: To minimize the risk of AEs, the investigators will monitor carefully to determine whether or not they are within the expected range. The degree of AEs is evaluated according to The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v 4.0). Investigators will also conduct a thorough examination and adopt an appropriate system to take any necessary measures to deal with AEs.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical study; fully understands and is informed of the study and has signed the Informed Consent Form (ICF).
2. The gender is not limited. Age: ≥ 18 years and ≤ 75 years old.
3. Gastric or gastroesophageal junction adenocarcinoma confirmed by pathology.
4. Without evidence of distant metastatic disease before operation by imaging.
5. Received D2 or D2+ radical gastrectomy by open surgery (R0 resection).
6. Stage III gastric cancer confirmed by postoperative pathology (AJCC/UICC 8th TNM staging classification).
7. Participants with a performance status of 0 ~ 1 on the Eastern Cooperative Oncology Group (ECOG) within 7 days before the first dose of study treatment.
8. Life expectancy ≥ 6 months.
9. The functions of the vital organs meet requirements as follow (within 14 days before the first dose of study treatment, participant has not received treatment of blood transfusion, albumin, recombinant human thrombopoietin or granulocyte stimulating factor):

   A. Hematological function：
   * White blood cell count (WBC): 3.5 × 10 ^ 9 / L ~12.0 × 10 ^ 9 / L；
   * Absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L；
   * Platelet count (PLT) ≥ 100 × 10 ^ 9 / L；
   * Hemoglobin (Hb) ≥ 90 g / L.

   B. Hepatic function：
   * Total bilirubin (TBIL) ≤ 1.5 × ULN (upper limit of normal);
   * Aspartate aminotransferase (AST) ≤ 2.5 × ULN;
   * Alanine aminotransferase (ALT) ≤ 2.5 × ULN;
   * Albumin (ALB) ≥ 30 g / L.

   C. Renal function：
   * Creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 60 ml / min for those with creatinine level > 1.5 × ULN.

   D. Coagulation function：
   * International normalized ratio (INR) ≤ 1.5;
   * Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
10. Female of childbearing age must meet requirements: urine pregnancy test must be negative within 7 days before the first dose of study treatment, and she must agree to use adequate contraception methods or keep abstinence (starting with the ICF is signed through 120 days after the last dose of camrelizumab, or 180 days after the last dose of chemotherapy, whichever is longer, and should not be breastfeeding. For the male participants must meet requirements: agree to use adequate contraception methods or keep abstinence (starting with the ICF is signed through 120 days after the last dose of camrelizumab, or 180 days after the last dose of chemotherapy, whichever is longer).

Exclusion Criteria:

1. Received previous chemotherapy, radiotherapy, targeted therapy or immunotherapy.
2. Previous or concurrent have other active malignant tumors (except for basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate cancer or cervical cancer or breast cancer in situ that has undergone curative therapy).
3. Existence of unrecovered complications after radical gastrectomy before the first dose of study treatment (including but not limited to: infection, gastrointestinal bleeding/ obstruction, anastomotic fistula, pancreatic fistula and anastomotic stenosis).
4. Myocardial infarction within 6 months before the first dose of study treatment, uncontrolled angina, arrhythmia which need medical intervention (including but not limited to cardiac pacemaker), congestive heart failure (New York Heart Association (NYHA) class III or IV), echocardiogram shows left ventricular ejection fraction (LVEF) < 50%.
5. Existence of chronic diarrhea (watery diarrhea: ≥ 5 times per day).
6. Participants with active infection within 14 days before the first dose of study treatment which need medical intervention.
7. Participants with active tuberculosis.
8. Previous or concurrent diagnosed with interstitial lung disease by imaging or symptoms.
9. Any of the following test is positive: Human Immunodeficiency Virus (HIV) antibody, Hepatitis B surface Antigen (HBsAg), or Hepatitis C Virus (HCV) antibody.
10. Females who are pregnant or breastfeeding or expecting to conceive during the study period.
11. Participants who need long-term systemic steroid therapy (> 10 mg/d prednisone equivalent) or any other form of immunosuppressive therapy within 14 days before the first dose of study treatment or during the study period.
12. Concurrent or previous have severe allergic reaction to any antibody-based drugs.
13. Existence of any concurrent autoimmune disease, excepting participants with diabetes mellitus type I, hypothyroidism requiring only hormone replacement therapy and skin diseases without systemic treatment (such as vitiligo, psoriasis or alopecia).
14. Receive live vaccines within 28 days before the first dose of study treatment or during the study period, excepting inactivated viral vaccines for seasonal influenza.
15. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
16. Existence of systemic disease that is difficult to control despite treatment with several agents, for example, diabetes mellitus, hypertension, etc.
17. Existence of other serious physical or mental diseases or serious laboratory abnormalities that may increase the risk of participating in the study. Participants who were judged unsuitable as subjects of this trial by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2026-03-29 (Estimated)

PRIMARY OUTCOMES:
The incidences and types of adverse events | 9 months
  The incidences and types of adverse events that occur during treatment will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  Disease-free survival (DFS)
Overall survival (OS) | 3 years
  Overall survival (OS)
Treatment completion rate | 6 months
  Percentage of participants who complete eight cycles of chemotherapy in combination with Camrelizumab.

CONTACTS AND LOCATIONS:
Overall Officials: Jiren Yu, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (4):
- China (4):
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Jin H, Yu J, Gao Y, Liu X, Xu H, Jiang H, Zhou S, Xu N, Zheng Y, Shen Q, Zhao Z, Wu D, Zhang Q, Zhu K. Camrelizumab plus SOX chemotherapy as adjuvant therapy for pathological stage III gastric or gastroesophageal junction adenocarcinoma: a prospective, multicenter, single-arm, phase II trial. Ther Adv Med Oncol. 2025 Jul 10;17:17588359251355781. doi: 10.1177/17588359251355781. eCollection 2025. PMID 40656603